CLINICAL TRIAL: NCT03288662
Title: Evaluate the Relationship Between Computed Tomography Manifestation and Histopathological Classification of Thymic Epithelial Tumors
Brief Title: Relationship Between Computed Tomography Manifestation and Histopathological Classification of Thymic Epithelial Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Military Hospital 103 (Other)
Collaborators: Nguyen Truong Giang (Unknown)
Responsible Party: Principal Investigator, Le Viet Anh, MD, Principal Investigator, Military Hospital 103
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LAnh
Record Dates: First submitted 2017-09-07; First posted 2017-09-20 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Thymoma
Keywords: Computed tomography; thymic epithelial tumors
MeSH Terms: conditions — Thymoma

STUDY DESIGN:
Intervention Model Description: Cross-sectional descriptive study on 53 patients with diagnosed of thymoma by CT and had postoperative histopathology results as thymic epithelial tumors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT and histopathological classification (Experimental): With each histopathological type of thymic epithelial tumors, we measure the maximun diameter in chest CT scan. Comparison of some characteristics of the tumor on preoperative chest CT scans and histopathological type of thymic epithelial tumors .
  Interventions: Other: CT and histopathological classification

INTERVENTIONS:
Other: CT and histopathological classification — Cross-sectional descriptive study on 53 patients with diagnosed of thymoma by CT and had postoperative histopathology results as thymic epithelial tumors. Base on the characteristics in Chest CT scan in each postoperative histopathology results.

SUMMARY:
the World Health Organization (WHO) has proposed a classification of histopathological thymic tumor and it significance in prognosis. Chest computed tomography (CT) is the most common method to evaluate thymic epithelial tumors before operation. Therefore, the question is to predict the histopathological type of thymic epithelial tumors before surgery based on CT-scan images , to help determine treatment strategy and prognosis. In Vietnam, there are no published literature on this issue.

DETAILED DESCRIPTION:
1. Introduction: the World Health Organization (WHO) has proposed a classification of histopathological thymic tumor and it significance in prognosis. Chest computed tomography (CT) is the most common method to evaluate thymic epithelial tumors before operation. Therefore, the question is to predict the histopathological type of thymic epithelial tumors before surgery based on CT-scan images , to help determine treatment strategy and prognosis. In Vietnam, there are no published literature on this issue.
2. Materials and methods:

   2.1. Cross-sectional descriptive study on 53 patients with diagnosed of thymoma by CT and had postoperative histopathology results as thymic epithelial tumors

   2.2. Time and Place: in Departement of CTVS, Military Hospital 103, Vietnam from 10/2013 to 7/2017.

   2.3. methods:
   * study in chest CT scan:

     * Measure the maximun diameter of the tumor
     * The contour: smooth contour or irregular contour
     * The shape: round, oval and plaque base on the ratio between long axis and short axis of the tumor
     * Some other characteristics: Degree of enhancement, Level of drug absorbed, Calcification, Invasion the local organs and Capsular destruction.
   * Histopathological study: based on the 2004 WHO classification:

     * Thymoma: type A, AB, B1, B2, B3
     * Thymic carcinoma
   * Data processing: use software Epi Info 2000.
3. Expectation of results

   * Relationship between the size and histopathological type of thymic epithelial tumors.
   * Comparison of some characteristics of the tumor on preoperative chest CT scans and histopathological type of thymic epithelial tumors

ELIGIBILITY:
Inclusion Criteria:

* All of patient have a chest CT scan pre-operation and a result of thymic epithelial tumors postoperative histopathology

Exclusion Criteria:

* Incomplete or loss the CT and postoperative histopathology

Ages: 21 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
maximun diameter of the tumor | 1 month
  Measure the maximun diameter of the tumor in chest CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Truong Giang Nguyen, PhD, Study Chair — VMMU

IPD SHARING:
Plan to Share IPD: Undecided